CLINICAL TRIAL: NCT03628924
Title: A Phase 2, Multicenter, Randomized, Placebo-Controlled, Double-Blind, Proof-of-Concept Study to Evaluate Guselkumab for the Treatment of Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of Guselkumab for the Treatment of Participants With Moderate to Severe Hidradenitis Suppurativa (HS)
Acronym: NOVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108500; 2018-001176-38 (EudraCT Number); CNTO1959HDS2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Guselkumab Regimen 1 (Experimental): Participants will receive guselkumab dose 1 administered Intravenously (IV) followed by guselkumab dose 2 administered subcutaneously.
  Interventions: Drug: Guselkumab dose 1; Drug: Guselkumab dose 2; Drug: Placebo
- Group 2: Guselkumab Regimen 2 (Experimental): Participants will receive guselkumab dose 2 subcutaneously.
  Interventions: Drug: Guselkumab dose 2; Drug: Placebo
- Group 3: Placebo then Guselkumab (Experimental): Participants will receive placebo IV and SC and an additional SC placebo dose at Week 12 then cross over at Week 16 to receive guselkumab dose 2 and dose 3 SC and placebo SC.
  Interventions: Drug: Guselkumab dose 2; Drug: Guselkumab dose 3; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab dose 1 — Participants will receive guselkumab dose 1 IV.
  Other Names: CNTO 1959
  Arms: Group 1: Guselkumab Regimen 1
Drug: Guselkumab dose 2 — Participants will receive guselkumab dose 2 SC in Group 1, 2 and Group 3.
  Other Names: CNTO 1959
Drug: Guselkumab dose 3 — Participants will receive guselkumab dose 3 SC in Group 3.
  Other Names: CNTO 1959
  Arms: Group 3: Placebo then Guselkumab
Drug: Placebo — Participants will receive matched placebo SC and IV in group 1, 2 and 3 with an additional placebo SC dose in Group 3.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of guselkumab in adult participants with moderate to severe hidradenitis suppurativa (HS).

ELIGIBILITY:
Inclusion Criteria:

* Have moderate to severe Hidradenitis Suppurativa (HS) for at least 1 year (365 days) prior to the baseline visit as determined by the investigator through participant interview and/or review of the medical history
* Have HS lesions present in at least 2 distinct anatomic areas (examples include but are not limited to left and right axilla; or left axilla and left inguinocrural fold)
* Had an inadequate response to an adequate course of appropriate oral antibiotics for treatment of HS (or demonstrated intolerance to, or had a contraindication to oral antibiotics for treatment of their HS) in the investigator's opinion
* Have a total abscess and inflammatory nodule (AN) count of greater than or equal to (>=) 3 at the screening and baseline visit
* Must agree to daily use (throughout the entirety of the study) of one of the following over-the-counter treatments to the body areas affected with HS lesions: either soap and water, or a topical antiseptic wash containing chlorhexidine gluconate, triclosan, or benzoyl peroxide, or a dilute bleach bath

Exclusion Criteria:

* Any other active skin disease or condition (example, bacterial, fungal or viral infection) that could have interfered with assessment of HS
* Has a draining fistula count of greater than (>) 20 at the baseline visit
* Receipt of prescription topical therapies for the treatment of HS within 14 days prior to the baseline visit
* Receipt of systemic non-biologic therapies for the treatment of HS less than (<) 4 Weeks prior to the baseline visit
* Receipt of any oral antibiotic treatment for HS or inflammatory disorders within 4 Weeks prior to the baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (45):
- United States (20):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Olympian Clinical Research, Largo, Florida
  - Renstar Medical Research, Ocala, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Forcare Clinical Research Inc, Tampa, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Indiana Clinical Trial Center, Plainfield, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Central Dermatology, St Louis, Missouri
  - Clinical Studies Group, Henderson, Nevada
  - Ohio State University, Columbus, Ohio
  - Oregon Medical Research Center, Portland, Oregon
  - University of Pittsburgh Department of Dermatology, Pittsburgh, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Progressive Clinical Research, San Antonio, Texas
  - Dermatology Associates of Seattle, Seattle, Washington
- Canada (4):
  - Dr Wei Jing Loo Medicine Professional Corporation, London, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
- Denmark (2):
  - Bispebjerg Hospital, København NV
  - Sjaellands University Hospital, Roskilde
- France (7):
  - Hopital Prive d'Antony, Antony
  - Groupe Hospitalier La Rochelle - Re - Aunis, La Rochelle
  - CHU de Nice, Nice
  - Polyclinique de Courlancy, Reims
  - Hopital Charles Nicolle, Rouen
  - CHU Saint Etienne, Saint-Priest-en-Jarez
  - Hopital Larrey CHU de Toulouse, Toulouse
- Germany (9):
  - Charite - Universitaetsmedizin Berlin (CCM), Berlin
  - Katholisches Klinikum Bochum gGmbH, Bochum
  - Klinikum Darmstadt GmbH - Hautklinik, Darmstadt
  - Stadtisches Klinikum Dresden, Dresden
  - Universitaetsklinik Erlangen, Erlangen
  - Universitatsklinikum Frankfurt, Frankfurt
  - Haut- und Laserzentrum Freising, Freising
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsmedizin Mainz, Mainz
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Radboudumc, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam

REFERENCES:
- [Derived] Kimball AB, Podda M, Alavi A, Miller M, Shen YK, Li S, Xu Y, Han C, Fakharzadeh S, Yang YW, DePrimo S, Munoz E, Chen Y, Passeron T, Papp K. Guselkumab for the treatment of patients with moderate-to-severe hidradenitis suppurativa: A phase 2 randomized study. J Eur Acad Dermatol Venereol. 2023 Oct;37(10):2098-2108. doi: 10.1111/jdv.19252. Epub 2023 Jun 27. PMID 37317022

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 184 enrolled participants, 181 participants received treatment. 3 participants were randomized but did not receive treatment.
Groups:
- Placebo (Week 0 - 16): Participants received placebo intravenously (IV) and subcutaneously (SC) at Weeks 0, 4, 8 and an additional SC placebo at Week 12.
- Guselkumab 200 Milligrams (mg) SC (Week 0 - 16): Participants received 200 mg guselkumab SC at Weeks 0, 4, 8, and 12.
- Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16): Participants received 1200 mg guselkumab IV at Weeks 0, 4, and 8, and 200 mg guselkumab SC at Week 12.
- Placebo Crossover to Guselkumab 100 mg SC (Week 16 - 48): At Week 16, participants receiving placebo during placebo-controlled period were re-randomized to receive 100 mg guselkumab SC at Weeks 16, 20, 28 and 36 and placebo at Weeks 24 and 32. All participants entered safety follow-up at Week 36 through Week 48.
- Placebo Crossover to Guselkumab 200 mg SC (Week 16 - 48): At Week 16, participants receiving placebo during placebo-controlled period were re-randomized to receive 200 mg guselkumab SC every 4 weeks (q4w) through Week 36. All participants entered safety follow-up at Week 36 through Week 48.
- Guselkumab 200 mg SC (Week 16 - 48): Participants who were receiving 200 mg guselkumab SC during placebo-controlled period, continued to receive 200 mg guselkumab SC q4w through Week 36. All participants entered safety follow-up at Week 36 through Week 48.
- Guselkumab 1200 mg IV Crossover to Guselkumab 200 mg SC (Week 16 - 48): Participants who were receiving 1200 mg guselkumab IV during placebo-controlled period switched treatment at Week 12 to receive guselkumab 200 mg SC q4w through Week 36. All participants entered safety follow-up at Week 36 through Week 48.
Period: Placebo Controlled Period (Week 0 - 16)
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16) | Placebo Crossover to Guselkumab 100 mg SC (Week 16 - 48) | Placebo Crossover to Guselkumab 200 mg SC (Week 16 - 48) | Guselkumab 200 mg SC (Week 16 - 48) | Guselkumab 1200 mg IV Crossover to Guselkumab 200 mg SC (Week 16 - 48)
Started | 62 | 59 | 60 | 0 | 0 | 0 | 0
Completed | 56 | 56 | 57 | 0 | 0 | 0 | 0
Not Completed | 6 | 3 | 3 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 1 | 0 | 0 | 0 | 0
Period: Active Treatment Period (Week 16-48)
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16) | Placebo Crossover to Guselkumab 100 mg SC (Week 16 - 48) | Placebo Crossover to Guselkumab 200 mg SC (Week 16 - 48) | Guselkumab 200 mg SC (Week 16 - 48) | Guselkumab 1200 mg IV Crossover to Guselkumab 200 mg SC (Week 16 - 48)
Started | 0 | 0 | 0 | 28 | 28 | 56 | 57
Completed | 0 | 0 | 0 | 20 | 24 | 43 | 46
Not Completed | 0 | 0 | 0 | 8 | 4 | 13 | 11
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 2 | 4
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 5 | 1 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16) | Total
Number analyzed (Participants) | 62 | 59 | 60 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 57 | 60 | 177
  >=65 years | 2 | 2 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (11.55) | 39 (12.37) | 37.2 (10.92) | 38.1 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 32 | 45 | 115
  Male | 24 | 27 | 15 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 6 | 17
  White | 46 | 42 | 43 | 131
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 6 | 13 | 11 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  CANADA | 8 | 8 | 6 | 22
  DENMARK | 2 | 0 | 2 | 4
  FRANCE | 13 | 18 | 20 | 51
  GERMANY | 13 | 13 | 10 | 36
  NETHERLANDS | 3 | 1 | 3 | 7
  UNITED STATES | 23 | 19 | 19 | 61

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 16
Description: HiSCR is defined as at least 50 percent (%) reduction in total abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count relative to baseline.
Time Frame: Week 16
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study intervention. Participants with missing data after applying treatment failure rules were assumed to be non-responders. Participants who discontinued study intervention due to lack of efficacy or Adverse event (AE) of worsening of hidradenitis suppurativa (HS), or who started protocol-prohibited medication or therapy during study that could improve HS were considered treatment failures.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 62 | 59 | 60
percentage of participants | 38.7 | 50.8 | 45.0
Statistical Analysis 1: Comparison: Placebo (Week 0 - 16) vs Guselkumab 200 Milligrams (mg) SC (Week 0 - 16); Test type: Superiority; p = 0.166, Cochran-Mantel-Haenszel; Treatment difference = 12.6, 95% CI 2-sided [-4.6 to 29.8]
Statistical Analysis 2: Comparison: Placebo (Week 0 - 16) vs Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16); Test type: Superiority; p = 0.459, Cochran-Mantel-Haenszel; Treatment difference = 6.6, 95% CI 2-sided [-10.3 to 23.6]

2. Secondary Outcome: Change From Baseline in Participant's Total Abscess and Inflammatory Nodule (AN) Count at Week 16
Description: Change from baseline in total AN count at Week 16 was reported. Abscess and inflammatory nodule were counted for the HS affected anatomical regions. The AN count is the sum of number of abscess and inflammatory nodules across anatomical regions.
Time Frame: Baseline and Week 16
Population: FAS included all randomized participants who received at least one administration of study intervention. The analysis was based on observed data after applying treatment failure rules (the change from baseline using observed data or 0 [no improvement] if a participant met treatment failure [TF] criteria). Here, N (number of participants analyzed) signifies participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: count of abscess and inflammatory nodule
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 59 | 57 | 59
count of abscess and inflammatory nodule | -3.2 (7.37) | -5.3 (9.29) | -5.3 (6.53)

3. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Week 16
Description: DLQI is a simple, compact, and practical questionnaire to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. The participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). The DLQI total score is derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best. A lower score (that is, negative change score) indicates improvement in the Quality of Life.
Time Frame: Baseline and Week 16
Population: FAS included all randomized participants who received at least one administration of study intervention. The analysis was based on observed data after applying treatment failure rules (the change from baseline using observed data or 0 [no improvement] if a participant met TF criteria). Here, N (number of participants analyzed) signifies participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 59 | 56 | 57
units on a scale | -0.7 (5.17) | -3.4 (6.81) | -2.5 (6.13)

4. Secondary Outcome: Change From Baseline in Hidradenitis Suppurativa (HS)-Related Pain Symptom Score in the Past 24 Hours Based on Hidradenitis Suppurativa Symptom Diary (HSSD) Questionnaire at Week 16
Description: HSSD is a 7-item patient self-reported questionnaire that assesses 5 HS-related symptoms including pain, tenderness, hot skin feeling, odor, and itchiness. The participants were asked to rate the severity of each symptom on a 0 to 10 numerical rating scale, with 0 indicating no symptom experience and 10 indicating the worst possible symptom experience. All 5 symptoms have a recall period of the past 7 days, except for 2 additional questions on pain which evaluate current pain and pain in the past 24 hours with a score range from 0 (no symptom experience) to 10 (worst possible symptom experience). A total symptom score also ranged from 0 (no symptom) to 10 (worst possible symptom), was derived by averaging the 5 individual scale scores that utilize the past 7-day recall period. Change from baseline in HS-related pain symptom score based on HSSD was reported.
Time Frame: Baseline and Week 16
Population: FAS included all randomized participants who received at least one administration of study intervention. Participants who received analgesic therapy for HS within 1 day of a scheduled visit date, the participants were considered a treatment failure at that visit (the change from baseline using observed data or 0 [no improvement] if a participant met TF criteria). Here, N (number of participants analyzed) signifies participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 56 | 55 | 56
units on a scale | -0.3 (3.17) | -1.6 (3.05) | -1.2 (2.93)

5. Secondary Outcome: Percentage of Participants Who Achieved at Least 50 Percent Reduction in Total Abscess and Inflammatory Nodule Count at Week 16
Description: Percentage of participants who achieved at least 50 percent reduction in total AN count at Week 16 were reported. Abscess and inflammatory nodule were counted for the HS affected anatomical regions. The AN count is the sum of number of abscess and inflammatory nodules across anatomical regions.
Time Frame: Week 16
Population: FAS included all randomized participants who receive at least one administration of study intervention. Participants with missing data after applying treatment failure rules were assumed to be non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 62 | 59 | 60
percentage of participants | 45.2 | 55.9 | 51.7

6. Secondary Outcome: Percentage of Participants Who Achieved at Least 75 Percent Reduction in Total Abscess and Inflammatory Nodule Count at Week 16
Description: Percentage of participants who achieved at least 75 percent reduction in total AN count at Week 16 were reported. Abscess and inflammatory nodule were counted for the HS affected anatomical regions. The AN count is the sum of number of abscess and inflammatory nodules across anatomical regions.
Time Frame: Week 16
Population: FAS included all randomized participants who received at least one administration of study intervention. Participants with missing data after applying treatment failure rules were assumed to be non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 62 | 59 | 60
percentage of participants | 30.6 | 40.7 | 26.7

7. Secondary Outcome: Percentage of Participants Who Achieved at Least 90 Percent Reduction in Total Abscess and Inflammatory Nodule Count at Week 16
Description: Percentage of participants who achieved at least 90 percent reduction in total AN count at Week 16 were reported. Abscess and inflammatory nodule were counted for the HS affected anatomical regions. The AN count is the sum of number of abscess and inflammatory nodules across anatomical regions.
Time Frame: Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 62 | 59 | 60
percentage of participants | 17.7 | 22.0 | 15.0

8. Secondary Outcome: Percentage of Participants Who Achieved 100 Percent Reduction in Total Abscess and Inflammatory Nodule Count at Week 16
Description: Percentage of participants who achieved 100 percent reduction in total AN count at Week 16 were reported. Abscess and inflammatory nodule were counted for the HS affected anatomical regions. The AN count is the sum of number of abscess and inflammatory nodules across anatomical regions.
Time Frame: Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 62 | 59 | 60
percentage of participants | 14.5 | 15.3 | 15.0

9. Secondary Outcome: Percentage of Participants Who Achieved an Abscess and Inflammatory Nodule Count of 0/1 and AN Count of 0/1/2 at Week 16
Description: Percentage of participants who achieved an AN count of 0/1 and AN Count of 0/1/2 at Week 16 were reported. Abscess and inflammatory nodule were counted for the HS affected anatomical regions. The AN count is the sum of number of abscess and inflammatory nodules across anatomical regions.
Time Frame: Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 62 | 59 | 60
percentage of participants
  AN Count of 0/1 | 27.4 | 30.5 | 23.3
  AN Count of 0/1/2 | 33.9 | 39.0 | 31.7

10. Secondary Outcome: Percentage of Participants Who Achieved Abscess Count of 0 at Week 16 For Participants With Baseline Abscess Count Greater Than 0
Description: Percentage of participants who achieved abscess count of 0 at Week 16 for participants with baseline abscess count greater than (>) 0 were reported.
Time Frame: Week 16
Population: Population analyzed included FAS participants with baseline abscess count > 0. Participants with missing data after applying treatment failure rules were assumed to be non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 28 | 36 | 31
percentage of participants | 39.3 | 63.9 | 45.2

11. Secondary Outcome: Change From Baseline in the Number of Abscesses at Week 16
Description: Change from baseline in number of abscesses at Week 16 was reported.
Time Frame: Baseline and Week 16
Population: FAS included all randomized participants who received at least one administration of study intervention. The analysis was based on observed data after applying treatment failure rules (the change from baseline using observed data or 0 (no improvement) if a participant met TF criteria). Here, N (number of participants analyzed) signifies participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: abscess
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 59 | 57 | 59
abscess | -0.4 (2.72) | -2.1 (4.56) | -1.6 (3.90)

12. Secondary Outcome: Change From Baseline in HSSD Symptom Scale Total Score at Week 16
Description: HSSD is a 7-item patient self-reported questionnaire that assesses 5 HS-related symptoms including pain, tenderness, hot skin feeling, odor, and itchiness. The participants were asked to rate the severity of each symptom on a 0 to 10 numerical rating scale, with 0 indicating no symptom experience and 10 indicating the worst possible symptom experience. All 5 symptoms have a recall period of the past 7 days, except for 2 additional questions on pain which evaluate current pain and pain in the past 24 hours. A total symptom score, also ranged from 0 (no symptom) to 10 (worst possible symptom), was derived by averaging the 5 individual scale scores that utilize the past 7-day recall period.
Time Frame: Baseline and Week 16
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 59 | 56 | 57
units on a scale | -0.19 (2.124) | -1.71 (2.325) | -0.82 (2.148)

13. Secondary Outcome: Change From Baseline in HSSD Symptom Scale Score (Other Than Pain in the Past 24 Hours) at Week 16
Description: HSSD is a 7-item patient self-reported questionnaire that assesses 5 HS-related symptoms including pain, tenderness, hot skin feeling, odor, and itchiness. The participants were asked to rate the severity of each symptom on a 0 to 10 numerical rating scale, with 0 indicating no symptom experience and 10 indicating the worst possible symptom experience. All 5 symptoms have a recall period of the past 7 days, except for 2 additional questions on pain which evaluate current pain and pain in the past 24 hours. Change from baseline in each individual HSSD component scale (other than pain in the past 24 hours) tenderness, hot skin feeling, odor and itchiness symptom, pain, and current pain score (rated on a scale of 0 [no symptom experience] to 10 [worst possible symptom experience]) were reported.
Time Frame: Baseline and Week 16
Population: FAS included all randomized participants who received at least 1 dose of study intervention. Analysis was based on observed data after applying TF rules (change from baseline using observed data or 0 [no improvement] if a participant met TF criteria). Here, N (number of participants analyzed) signifies participants who were evaluated for this outcome measure and n (number of participants analyzed) signifies participants who were evaluated for this outcome measure for specified categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 59 | 56 | 57
units on a scale
  Change in HSSD Tenderness Scale Score | -0.4 (2.78) | -2.1 (2.93) | -1.3 (2.56)
  Change in HSSD Hot Skin Feeling Scale Score | 0.1 (2.85) | -1.6 (3.12) | -0.2 (3.16)
  Change in HSSD Odor Scale Score | -0.4 (2.73) | -1.9 (2.58) | -1.2 (2.77)
  Change in HSSD Itchiness Scale Score | 0.1 (2.82) | -1.1 (3.28) | -0.5 (2.85)
  Change in HSSD Pain Scale Score: number analyzed (Participants) | 56 | 55 | 56
  Change in HSSD Pain Scale Score | -0.3 (2.64) | -1.8 (2.86) | -0.9 (2.34)
  Change in HSSD Current Pain Score: number analyzed (Participants) | 56 | 55 | 56
  Change in HSSD Current Pain Score | -0.4 (2.71) | -1.5 (2.94) | -1.2 (2.76)

14. Secondary Outcome: Percentage of Participants Who Achieved Draining Fistula Count of 0 at Week 16 for Participants With Baseline Draining Fistula Count Greater Than 0
Description: Percentage of participants who achieved draining fistulas count of 0 at Week 16 for participants with baseline draining fistula count >0 were reported. Draining fistula were defined as fistulas that drain serous or purulent fluid, either spontaneously or by gentle palpation.
Time Frame: Week 16
Population: Population analyzed included FAS participants with baseline draining fistula count > 0. Participants with missing data after applying treatment failure rules were assumed to be non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 41 | 42 | 39
percentage of participants | 36.6 | 31.0 | 20.5

15. Secondary Outcome: Change From Baseline in Number of Draining Fistulas at Week 16
Description: Change from baseline in number of draining fistulas at Week 16 was reported. Draining fistula are defined as fistulas that drain serous or purulent fluid, either spontaneously or by gentle palpation.
Time Frame: Baseline and Week 16
Population: FAS included all randomized participants who received at least one administration of study intervention. The analysis was based on observed data after applying treatment failure rules (the change from baseline using observed data or 0 [no improvement] if a participant met TF criteria). Here, N (number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: fistulas
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 59 | 57 | 59
fistulas | -0.5 (2.87) | -1.7 (3.77) | -0.8 (2.08)

16. Secondary Outcome: Percentage of Participants Who Achieved Inflammatory Nodules Count of 0 at Week 16 for Participants With Baseline Inflammatory Nodule Count Greater Than 0
Description: Percentage of participants who achieved inflammatory nodules count of 0 at Week 16 in participants with baseline inflammatory nodules count >0 were reported.
Time Frame: Week 16
Population: Population analyzed included FAS participants with baseline inflammatory nodule count > 0. Participants with missing data after applying treatment failure rules were assumed to be non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 62 | 58 | 59
percentage of participants | 17.7 | 17.2 | 18.6

17. Secondary Outcome: Change From Baseline in Number of Inflammatory Nodules at Week 16
Description: Change from baseline in number of inflammatory nodules at Week 16 was reported.
Time Frame: Baseline and Week 16
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: inflammatory nodule
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 59 | 57 | 59
inflammatory nodule | -2.8 (6.96) | -3.2 (7.84) | -3.7 (4.91)

18. Secondary Outcome: Percentage of Participants With Hidradenitis Suppurativa-investigator's Global Assessment (HS-IGA) Score of Inactive (0), Almost Inactive (1), or Mild Activity (2) and With at Least 2-Grade Improvement Relative to Baseline at Week 16
Description: The HS-IGA documents the investigator's assessment of the participant's HS at a given timepoint. The anatomic region with the most severe HS activity at the baseline was evaluated for erythema, drainage, and pain and/or tenderness to palpation for each participant. The participant's HS is assessed as inactive (0), almost inactive (1), mild activity (2), moderate activity (3), or severe activity (4). A higher score indicates more severe disease. Percentage of participants with HS-IGA score of inactive (0), almost inactive (1), or mild activity (2) and with at least 2-grade improvement relative to baseline at Week 16 were reported.
Time Frame: Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 62 | 59 | 60
percentage of participants
  HS-IGA scores of inactive (0) | 16.1 | 13.6 | 13.3
  HS-IGA scores of inactive (0) or almost inactive (1) | 24.2 | 28.8 | 23.3
  HS-IGA scores of inactive (0), almost inactive (1), or mild activity (2) | 24.2 | 35.6 | 31.7

19. Secondary Outcome: Percentage of Participants With HS-IGA Score of Inactive (0) or Almost Inactive (1) at Week 16 Among Participants With HS-IGA Score of Moderate Activity (3) or Severe Activity (4) at Baseline
Description: The HS-IGA documents the investigator's assessment of the participant's HS at a given timepoint. The anatomic region with the most severe HS activity at the baseline was evaluated for erythema, drainage, and pain and/or tenderness to palpation for each participant. Among participants with score of moderate activity (3) or severe activity (4) at baseline, the same anatomic site selected for evaluation at the baseline were re-evaluated at Week 16. The participant's HS is assessed as inactive (0), almost inactive (1), mild activity (2), moderate activity (3), or severe activity (4). A higher score indicates more severe disease. Percentage of participants with HS-IGA score of inactive (0), almost inactive (1) at Week 16 among participants with HS-IGA score of moderate activity (3) or severe activity (4) at baseline were reported.
Time Frame: Week 16
Population: Population analyzed included FAS participants with HS-IGA scores of moderate activity (3) or severe activity (4) at baseline. Participants with missing data after applying treatment failure rules were assumed to be non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 55 | 49 | 52
percentage of participants | 27.3 | 32.7 | 25.0

20. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Total Score at Week 16
Description: The HADS has been developed to identify symptoms of anxiety and depression in hospitalized participants and in outpatients. It comprises 14 items, seven to assess anxiety (HADS-A), namely items 1, 3, 5, 7, 9, 11, and 13; and seven to assess depression (HADS-D), namely items 2, 4, 6, 8, 10, 12, and 14. Each item receives a score from 0 to 3 on a Likert Scale. The total score for each HADS-A and HADS-D scale is obtained by adding the individual scores for each item, with the maximum score 21. The presence or absence of depression and anxiety was defined, for each respective scale, based on the following cutoff values: HADS (anxiety): 0-8 equal to (=) no anxiety; greater than (>) 9 = anxiety; HADS (depression): 0-8 = no depression; >9 = depression.
Time Frame: Baseline and Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 59 | 57 | 57
units on a scale
  HADS-A | 0.0 (2.60) | 0.0 (2.82) | -0.3 (2.56)
  HADS-D | 0.2 (2.48) | -0.6 (2.73) | -0.5 (2.69)

21. Secondary Outcome: Change From Baseline in High-sensitivity C-Reactive Protein (Hs-CRP) at Week 16
Description: Change from baseline in hs-CRP at Week 16 was reported. Serum samples were collected and analyzed for hsCRP. Change from Baseline was calculated as: ([hs-CRP value at Week 16 minus Baseline value] divided by [Baseline value]).
Time Frame: Baseline and Week 16
Population: FAS included all randomized participants who received at least one administration of study intervention. Participants with missing data after applying treatment failure rules were assumed to be non-responders. Here, N (number of participants analyzed) signifies participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 52 | 51 | 52
milligrams per deciliter | -0.308 (8.0840) | 3.238 (19.0716) | -2.828 (11.1048)

22. Secondary Outcome: Number of Participants With Patient Global Impression of Change (PGIC) of Hidradenitis Suppurativa Severity Scale Score at Week 16
Description: The PGIC of HS Severity is a questionnaire that measures participants' perceived change (improvement or deterioration) in severity of their HS. Participants rated how his/her HS has changed since the beginning of the study using a 7-point scale ranging from 1 which indicates "a lot better now" to 7 which indicates "a lot worse now" with a neutral center point 4 which indicates ("neither better nor worse"). Participants' PGIC of HS Severity scale score at Week 16 were reported
Time Frame: Week 16
Population: FAS included all randomized participants who received at least one administration of study intervention. Participants with missing data after applying treatment failure rules are assumed to be 'Not improved'. Here, N (number of participants analyzed) signifies participants who were evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16)
Number analyzed (Participants) | 56 | 56 | 56
Participants
  A lot better now | 4 | 13 | 10
  Moderately better now | 7 | 14 | 11
  A little better now | 16 | 10 | 12
  No change | 20 | 12 | 18
  A little worse now | 3 | 2 | 4
  Moderately worse now | 5 | 1 | 1
  A lot worse now | 1 | 4 | 0

ADVERSE EVENTS:
Time Frame: Up to 48 weeks
Description: Safety analysis set included all participants who received at least 1 dose (complete or partial) of study intervention and participants were analyzed based on the treatment they actually received, regardless of the treatment groups to which they were assigned.
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16) | Placebo Crossover to Guselkumab 100 mg SC (Week 16 - 48) | Placebo Crossover to Guselkumab 200 mg SC (Week 16 - 48) | Guselkumab 200 mg SC (Week 16 - 48) | Guselkumab 1200 mg IV Crossover to Guselkumab 200 mg SC (Week 16 - 48)
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/59 | 0/60 | 0/28 | 0/28 | 0/56 | 0/57
Serious Adverse Events (participants affected / at risk) | 3/62 | 1/59 | 1/60 | 3/28 | 0/28 | 3/56 | 2/57
Other Adverse Events (participants affected / at risk) | 22/62 | 28/59 | 31/60 | 12/28 | 9/28 | 19/56 | 28/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0 - 16) (N=62) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) (N=59) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16) (N=60) | Placebo Crossover to Guselkumab 100 mg SC (Week 16 - 48) (N=28) | Placebo Crossover to Guselkumab 200 mg SC (Week 16 - 48) (N=28) | Guselkumab 200 mg SC (Week 16 - 48) (N=56) | Guselkumab 1200 mg IV Crossover to Guselkumab 200 mg SC (Week 16 - 48) (N=57)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small Intestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression Suicidal (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0 - 16) (N=62) | Guselkumab 200 Milligrams (mg) SC (Week 0 - 16) (N=59) | Guselkumab 1200 mg IV to Gus 200 mg SC (Week 0 - 16) (N=60) | Placebo Crossover to Guselkumab 100 mg SC (Week 16 - 48) (N=28) | Placebo Crossover to Guselkumab 200 mg SC (Week 16 - 48) (N=28) | Guselkumab 200 mg SC (Week 16 - 48) (N=56) | Guselkumab 1200 mg IV Crossover to Guselkumab 200 mg SC (Week 16 - 48) (N=57)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 1 | 3 | 0 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 6 | 0 | 0 | 4 | 1
Fatigue (General disorders) | 2 | 2 | 7 | 0 | 1 | 1 | 2
Oedema Peripheral (General disorders) | 0 | 1 | 2 | 2 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 4
Influenza (Infections and infestations) | 3 | 1 | 3 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 12 | 9 | 4 | 8 | 10 | 12
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 3 | 5 | 1 | 0 | 1 | 3
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 5 | 1 | 3 | 0 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 7 | 6 | 2 | 3 | 0 | 2 | 3
Migraine (Nervous system disorders) | 0 | 1 | 3 | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 1 | 0 | 1 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 3 | 7 | 2 | 4 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT03628924/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/24/NCT03628924/SAP_001.pdf